CLINICAL TRIAL: NCT06389942
Title: A Single-center, Randomized, Double-Blind, Placebo-Controlled Phase 1 Single Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity Characteristics of 9MW3011 in Healthy Volunteers
Brief Title: Single Ascending Dose Study of 9MW3011 in Chinese Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 9MW3011-2022-CP101
Record Dates: First submitted 2024-02-25; First posted 2024-04-29 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 9MW3011 Dose 1 (Experimental): Ascending IV doses administered per protocol
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo
- 9MW3011 Dose 2 (Experimental): Ascending IV doses administered per protocol
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo
- 9MW3011 Dose 3 (Experimental): Ascending IV doses administered per protocol
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo
- 9MW3011 Dose 4 (Experimental): Ascending IV doses administered per protocol
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo
- 9MW3011 Dose 5 (Experimental): Ascending IV doses administered per protocol
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo
- 9MW3011 Dose 6 (Experimental): Ascending IV doses administered per protocol
  Interventions: Drug: 9MW3011; Drug: 9MW3011 placebo

INTERVENTIONS:
Drug: 9MW3011 — Single dose intravenously on day 1
Drug: 9MW3011 placebo — Single dose intravenously on day 1

SUMMARY:
The objectives of the study are to evaluate the safety , tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of single ascending intravenous (IV) doses of 9MW3011 in Chinese healthy volunteers.

DETAILED DESCRIPTION:
The single ascending dose(SAD) study will comprise 6 dose cohorts of 8 healthy volunteers each. In each cohort, subjects will be randomized in a 6:2 ratio to receive 9MW3011 or placebo via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 65 years (including 18 and 65 years).
2. Weight≥50.0 kg for males, or weight≥45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 26.0 kg/m2 (including cut-off value).
3. Being judged by the investigator to be eligible based on medical history, physical examination, laboratory tests and test related items of inspection or no clinically significant mild abnormalities.
4. Volunteered to participate in this clinical trial, capable of giving written informed consent.

Exclusion Criteria:

1. Nervous/mental, respiratory system, cardiovascular system, digestive system, blood and lymphatic system, endocrine system, skeletal and muscular system , immune system, urinary system diseases , or a family history of severe systemic diseases (including cardiovascular system, digestive system, urinary system, etc.), may affect the health status of the subjects or any other diseases and physiological conditions that may affect the results of the study , judged by the investigator.
2. Currently suffering from iron deficiency/Iron deficiency anemia, taking iron supplements and complicated with other diseases related to abnormal iron metabolism.
3. Subjects who have a history of allergies to monoclonal antibodies or any drug components; those who have a history of allergies to excipients of 9MW3011.
4. Subjects who have lost blood or donated blood ≥200mL within 3 months before screening, or those who plan to donate blood within 3 months.
5. Positive for hepatitis B virus surface antigen and/or hepatitis B virus e antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, or treponema pallidum antibody.
6. Subjects who is inappropriate to participate in the trial due to any reasons as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Adverse Event(including serious adverse event) | up to day 99
  The incidence of AEs and SAEs from treatment until the last scheduled follow-up visit

SECONDARY OUTCOMES:
Number of subjects with abnormal vital signs | up to day 99
  Vital signs measurements will include pulse rate, respiration rate, blood pressure (systolic and diastolic blood pressure) and body temperature.
Number of subjects with abnormal clinically significant results from physical examination | up to day 99
  The physical examinations will include examination of the following: skin and mucous membranes, lymph nodes, head and neck, chest, abdomen, musculoskeletal, nervous system, and other sites of note elicited from the subject.
Number of subjects with abnormal clinically significant 12-lead electrocardiogram (ECG) parameters | up to day 99
  The examination indicators include heart rate, PR, QRS, uncorrected QT, and QTcF(corrected by Fridericia formula).
Number of subjects with abnormal clinically significant clinical laboratory results | up to day 99
  Clinical laboratory tests include hematology, urinalysis, blood chemistry, coagulation function.
Cmax | up to day 85
  The peak concentration
AUC0-t | up to day 85
  The area under the concentration-time curve from zero to the last time point
AUC0-∞ | up to day 85
  The area under the concentration-time curve from zero to infinity
Tmax | up to day 85
  The time to reach peak concentration
λz | up to day 85
  Terminal elimination rate constant
t1/2z | up to day 85
  The terminal elimination half-life
Vz | up to day 85
  The volume of distribution
CL | up to day 85
  Clearance
MRT | up to day 85
  Mean residence time
Pharmacodynamic(PD)parameters-hepcidin | up to day 85
  Change from baseline in hepcidin levels
PD parameters-serum iron | up to day 85
  Change from baseline in serum iron levels
PD parameters-TSAT | up to day 85
  Change from baseline in transferrin saturation(TSAT) levels
Anti-drug antibodies(ADA) | up to day 85
  The incidence of ADA

CONTACTS AND LOCATIONS:
Locations (1):
- PKUcare Luzhong Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: No